CLINICAL TRIAL: NCT04853797
Title: Effect of Ivabradine on Levcromakalim-Induced Symptoms in Individuals With Migraine Without Aura: A Randomized Double-Blind Two-Way Crossover Study
Brief Title: Effect of Ivabradine on Levcromakalim-Induced Symptoms in Individuals With Migraine Without Aura (ILIM)
Acronym: ILIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Ivabradine H-20061329
Record Dates: First submitted 2021-03-16; First posted 2021-04-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Headache; Migraine Without Aura
MeSH Terms: conditions — Headache; Migraine without Aura | interventions — Cromakalim; Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim - Ivabradine (Active Comparator): Infusion of levcromakalim (2.5 nmol minutes-1 over 20 minutes) followed by oral administration of ivabradine (15 mg orally).
  Interventions: Drug: Levcromakalim; Drug: Ivabradine
- Levcromakalim - Placebo (Placebo Comparator): Infusion of levcromakalim (2.5 nmol minutes-1 over 20 minutes) followed by oral administration of placebo.
  Interventions: Drug: Levcromakalim; Drug: Placebo

INTERVENTIONS:
Drug: Levcromakalim — 20 min infusion of 1 mg Levcromakalim followed by either oral Ivabradine or Placebo.
Drug: Ivabradine — 15 mg oral Ivabradine.
  Arms: Levcromakalim - Ivabradine
Drug: Placebo — Oral placebo (calcium supplements).
  Arms: Levcromakalim - Placebo

SUMMARY:
This study aims to explore the effect of Ivabradine on Levcromakalim-induced migraine in individuals with migraine without aura.

DETAILED DESCRIPTION:
Hyperpolarization-activated cation (HCN) channels have recently been implicated in neuropathic and inflammatory pain processes through their hyperfunction and/or overexpression.

HCN channels may play a significant role in migraine pathophysiology, as 1) both an inflammatory and a neuropathic component has been hypothesized to contribute to migraine, and 2) HCN channel activity is facilitated by cyclic nucleotides, e.g. cAMP and cGMP (molecules thought to be central in migraine pathophysiology) and increases in extracellular K+ concentration.

Opening of adenosine 5'-triphosphate-sensitive potassium channels (KATP channels) using Levcromakalim causes migraine attacks with and without aura in a high proportion of patients. KATP channel activation leads to hyperpolarization, which in turn could increase the open probability of HCN channels.

This study aims to explore the effects of Ivabradine on Levcromakalim-induced migraine in individuals with migraine without aura.

The investigators anticipate that this project will contribute greatly to the current understanding of migraine pathophysiology and the hypothesized role of HCN channels in migraine pain mechanisms. This is of great interest in future research, as such knowledge is an important prerequisite for further investigation and understanding of intracellular signalling mechanisms in migraine, which in turn will lead to the development of more effective and mechanism-based drugs.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give voluntary written informed consent to participate.
* Have a diagnosis of episodic migraine without aura according to The International Classification of Headache Disorders 3rd Edition.
* Be in good general health and without any cardio- or cerebrovascular diseases, psychiatric disorders or other severe comorbidities.
* Be 18-60 years of age.
* Have a weight between 50-100 kg.
* Have a normal standard resting 12-lead ECG at the screening visit with heart rate (HR) ≥ 60 bpm (the inclusion criterium of HR ≥ 60 bpm at screening has previously been used in studies with dosages of ivabradine up to 20 mg as single and multiple doses with no significant adverse events).
* Be without any chronic use of medicine.
* Have a negative urine-human chorionic gonadotropin (hCG) test at the screening visit if they are female of childbearing potential.

Exclusion Criteria:

* Suffer from tension type headache, as defined by the The International Classification of Headache Disorders 3rd Edition, more than five days a month on average in the last year.
* Are diagnosed with any primary headache disorder apart from migraine without aura as de-fined in The International Classification of Headache Disorders 3rd Edition (relating to tension type headache, see above).
* Suffer from any headache 48 hours prior to the start of the experiment or any migraine 72 hours prior to the start of the experiment.
* Are allergic to ivabradine or levcromakalim.
* Are lactose intolerant (due to Ivabradine tablets containing lactose).
* Have a daily intake of any medicine other than oral contraception or use of drugs or other ed-ibles/beverages with potential serious interactions with ivabradine
* Have a history of personal/familial or clinical signs of: cardiovascular and cerebrovascular disease (Long QT Syndrome, Cardiac dysrhythmia, Bradycardia, i.e. a resting heart rate of < 60 bpm at screening, Amnestic information or clinical signs of hyper- or hypotension (Hypertension (systolic blood pressure > 150 mmHg and / or diastolic blood pressure > 100 mmHg)/Hypotension (systolic blood pressure < 90 mm Hg and / or diastolic blood pressure < 50 mmHg)), Heart failure (NYHA II or higher)); Psychiatric conditions; Drug abuse of any kind; Smoking; Other comorbidities or clinical signs of diseases of any kind considered by the investigating physician to make the participant ineligible because of safety concerns).
* Are pregnant, breastfeeding or not using appropriate contraception.
* Do not want any information on significant pathological findings in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-07-06 (Actual)

PRIMARY OUTCOMES:
Incidence of migraine attacks | Assessed from baseline to 12 hours after infusion of levcromakalim
  A migraine attack is defined as an attack fulfilling either (i) or (ii):
  (i) Headache fulfilling criteria C and D for migraine without aura according to the International Headache Society criteria:
  C. Headache has at least two of the following characteristics:
  * unilateral location
  * pulsating quality
  * moderate or severe pain intensity (moderate to severe pain intensity is considered ≥4 on verbal rating scale)
  * aggravation by cough (in-hospital phase) or causing avoidance of routine physical activity (out-hospital phase)
  D. During headache at least one of the following:
  * nausea and/or vomiting
  * photophobia and phonophobia
  (ii) Headache described as mimicking the patient's usual migraine attack and treated with acute migraine medication (rescue medication).

SECONDARY OUTCOMES:
Incidence of headache | Assessed from baseline to 12 hours after infusion of levcromakalim
  Incidence of headache is defined as headache intensity ≥1 as measured by a numerical rating scale (NRS) from 0 to 10. It is a verbally declared scale from 0 to 10, where 0 is no pain; 10 is the worst pain imaginable
Intensity of headache | Assessed from baseline to 12 hours after infusion of levcromakalim
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no pain; 10 is the worst pain imaginable.
Changes in cerebral hemodynamics (velocity of blood flow in middle cerebral artery and diameter of superficial temporal artery) assessed using Transcranial Doppler Ultrasound (TCD) and high-frequency ultrasound (Dermascan C, Cortex Technology, Denmark) | Assessed from baseline until 150 minutes after levcromakalim infusion.
  Changes in cerebral hemodynamics will be assessed using Transcranial Doppler Ultrasound (TCD) (2 Mhz, DWL) to measure the velocity of middle cerebral artery (VMCA) blood flow bilaterally, and high-frequency ultrasound (Dermascan C, Cortex Technology, Denmark) to measure the diameter of the superficial temporal artery (STA) bilaterally.
Changes in blood pressure | Assessed from baseline until 150 minutes after levcromakalim infusion.
  Changes in blood pressure (systolic and diastolic) over time.
Heart rate | Assessed from baseline until 150 minutes after levcromakalim infusion.
  Changes in heart rate over time.
Incidence of adverse events | Assessed from baseline to 12 hours after infusion of Levcromakalim.
  Participants are instructed to inform the investigators in the case of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Prof., Principal Investigator — Danish Headache Center
Locations (2):
- Denmark (2):
  - Danish Headache Centre, Rigshospitalet-Glostrup, Glostrup, Region Sjælland
  - Danish Headache Center, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No